CLINICAL TRIAL: NCT04922190
Title: Promoting Physical Activity Engagement for People With Early-mid Stage Parkinson's Disease (Engage-PD)
Acronym: Engage-PD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-005
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: physical activity; exercise; rehabilitation
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Coaching (Experimental): Participants will receive up to 5 coaching sessions by a physical or occupational therapist. The intervention will focus on facilitating physical activity engagement and development of specific and measurable goals. The recommended program will be individualized to each participant but will primarily focus on increasing general physical activity (e.g. steps per day) as well as engagement in moderate intensity aerobic exercise a minimum of three times per week. At the follow up sessions the therapist will review progress with the current exercise plan and progress and discuss barriers and facilitators for exercise engagement. Participants will have the option to use a Fitbit or other device to monitor their heart rate and physical activity during the course of the intervention period.
  Interventions: Behavioral: Physical Activity Coaching

INTERVENTIONS:
Behavioral: Physical Activity Coaching — Participants will receive up to 5 coaching sessions by a physical or occupational therapist. The intervention will focus on facilitating physical activity engagement and development of specific and measurable goals. The recommended program will be individualized to each participant but will primarily focus on increasing general physical activity (e.g. steps per day) as well as engagement in moderate intensity aerobic exercise a minimum of three times per week. At the follow up sessions the therapist will review progress with the current exercise plan and progress and discuss barriers and facilitators for exercise engagement. Participants will have the option to use a Fitbit or other device to monitor their heart rate and physical activity during the course of the intervention period.

SUMMARY:
Engage-PD is a single cohort evaluation of implementation of a telehealth-delivered physical activity coaching program for people with early-mid stage Parkinson's disease. The program utilizes a physical or occupational therapist to provide one-on-one coaching for individuals with early-mid stage Parkinson's disease to provide individualized structured support to facilitate and optimize exercise uptake as part of an effective self-management program. The structure of the coaching program is based on previous research in neurodegenerative disease including Parkinson's disease and Huntington's disease.

DETAILED DESCRIPTION:
Individuals will be recruited through the Columbia University Medical Center Parkinson's Disease Center of Excellence. Individuals who choose to participate will first be given a brief evaluation, including history and contraindications for exercise, assessment of gait and balance, physical activity questionnaire (Brunel Lifestyle Inventory and International Physical Activity Questionnaire), pain questionnaire (Brief Pain Inventory), NeuroQOL quality of life assessment, and a self-efficacy measure about exercise engagement (Exercise Self Efficacy Scale). For those individuals who report low back pain, we will further administer the Modified Oswestry Low Back Pain Disability Questionnaire and a customized low back pain questionnaire. The therapist will then conduct the coaching session (see below). If this assessment is not able to be conducted in person, it will be conducted via secure videoconferencing. There will be between 1-4 follow-up phone call/videosessions and a follow-up assessments at 3 months and 6 months where all assessment will be repeated. A short questionnaire will also be administered at 3 and 6 months to assess the acceptability of the intervention.

The coaching program will utilize the Pre-Active PD program (Clinicaltrials.gov NCT03696589) to guide the delivery of the intervention. This will include a checklist of the key elements that are important for the therapist in order to facilitate PA behavior change. In addition, the therapist will utilize motivational interviewing strategies that include four processes (engaging, evoking, planning, and tracking) and five core communication skills (asking open ended questions, affirming, reflective listening, summarizing, and informing and advising). The therapist will introduce the Pre-Active PD workbook and utilize it as a tool and reference for the participant in order to engage and focus them throughout the coaching process, and will educate participants on the types of exercise options and the specific exercise benefits for PD. In the planning process, the therapist will facilitate discussion on development of specific and measurable goals, and will provide options for tracking their progress, such as written or web-based exercise logs or an activity monitor. The recommended exercises will be individualized to each participant but will primarily focus on increasing general physical activity (e.g. steps per day) as well as engagement in moderate-vigorous intensity aerobic exercise a minimum of three times per week. Balance and strengthening exercises will also be recommended as appropriate. At the follow up sessions (15-30 min), the therapist will review progress with the current exercise plan and progress, record if any falls have occurred and discuss barriers and facilitators for exercise engagement. Participants will also be given a short exercise safety checklist to assure safety when conducting home exercises. Participants will have the option to use a Fitbit device (Charge 4) to monitor their heart rate and physical activity during the course of the intervention period. Participants will use a study-specific login to track their progress and activity. Participants who already own a Fitbit or other activity monitor can continue to use their device during the study.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist confirmed clinical diagnosis for Parkinson's disease Hoehn & Yahr stage I-III
* Ambulatory for indoor and outdoor mobility without assistance or assistive device
* Successful completion of Physical Activity Readiness Questionnaire (PAR-Q)26 or medical clearance from GP

Exclusion Criteria:

* Musculoskeletal injury that would prevent participation in an exercise program
* Other neurological disease or disorder such as stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Brunel Lifestyle Physical Activity Questionnaire | 3 months
  The Brunel lifestyle inventory is a 10-item questionnaire that measures both pre-planned (6 items) and un-planned (3 items) lifestyle PA. Scoring for each item is on a scale of 1-5, and the scores for each subscale are averaged. Scores range from 1 (low level of physical activity) to 5 (high level of physical activity).
Self-Efficacy for Exercise Scale | 3 months
  18-item test that measures an individual's self-efficacy to participate in exercise when numerous barriers are present, including both social and physical barriers. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (Short-Form Phone version) | 3 months
  Evaluates physical activity over the previous 7 days represented in MET/min per week with higher values meaning greater physical activity.
NeuroQOL | 3 months
  Patient-reported questionnaire evaluating sleep disturbances, depression, fatigue and social participation and satisfaction.
Brief Pain Inventory | 3 months
  Evaluates the presence of pain including intensity and interference with activities of daily living. Mean of the four severity items is used as measures of pain severity; the mean of the seven interference items is used as a measure of pain interference.
Timed Up and Go | 3 months
  Performance-based assessment which requires a person to stand up from a chair, walk 10 feet, turn around, return to their chair and sit back down. Outcome is measured in time (sec) to complete and higher value is worse performance.
Standing balance assessment | 3 months
  Participant will perform static standing with feet together and postural sway will be recorded with a smartphone app.
Modified Oswestry Low Back Pain Disability Questionnaire | 3 months
  Questionnaire evaluating how back pain affects everyday life (optional for those participants who report low back pain). Range 0-50 with 50 being higher level of disability.
Acceptability questionnaire (open-ended questions) | 3 months
  A short open-ended questionnaire to assess the acceptability of the intervention. These open-ended questions will be analyzed qualitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No